CLINICAL TRIAL: NCT02685462
Title: A Phase 1 Open-Label Study in Healthy Adult Subjects to Assess the Effect of Cenicriviroc Mesylate (CVC) on the Pharmacokinetics (PK) of HMG-CoA Reductase Inhibitors (Rosuvastatin, Atorvastatin and Simvastatin), Caffeine and Digoxin
Brief Title: Pharmacokinetic and Safety Study of Cenicriviroc and HMG-CoA Reductase Inhibitors, Caffeine and Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 652-124
Record Dates: First submitted 2016-02-03; First posted 2016-02-18 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Atorvastatin; Simvastatin; Digoxin; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Rosuvastatin) (Active Comparator): Group 1 (12 subjects) will receive Rosuvastatin on Days 1 and 13.
  Interventions: Drug: Rosuvastatin
- Group 1 (Digoxin) (Active Comparator): Group 1 (12 subjects) will receive Digoxin on Days 1 and 13.
  Interventions: Drug: Digoxin
- Group 1 (Caffeine) (Active Comparator): Group 1 (12 subjects) will receive Caffeine on Days 1 and 13.
  Interventions: Drug: Caffeine
- Group 2 (Atorvastatin) (Active Comparator): Group 2 (12 subjects) will receive Atorvastatin on Days 1 and 13.
  Interventions: Drug: Atorvastatin
- Cenicriviroc (Experimental): Subjects in Group 1 and Group 2 will receive Cenicriviroc on Days 3-12.
  Subjects in Group 3 will receive Cenicriviroc on Days 2-12.
  Interventions: Drug: Rosuvastatin; Drug: Atorvastatin; Drug: Simvastatin; Drug: Digoxin; Drug: Caffeine
- Group 3 (Simvastatin) (Active Comparator): Group 3 (12 subjects) will receive Simvastatin on Days 1 and 12.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Rosuvastatin 20 mg
  Arms: Cenicriviroc; Group 1 (Rosuvastatin)
Drug: Atorvastatin
  Other Names: Atorvastatin 20 mg
  Arms: Cenicriviroc; Group 2 (Atorvastatin)
Drug: Simvastatin
  Other Names: Simvastatin 20 mg
  Arms: Cenicriviroc; Group 3 (Simvastatin)
Drug: Digoxin
  Other Names: Digoxin 0.25 mg
  Arms: Cenicriviroc; Group 1 (Digoxin)
Drug: Caffeine
  Other Names: Caffine 200 mg
  Arms: Cenicriviroc; Group 1 (Caffeine)

SUMMARY:
This is a Phase 1, Open-Label, 3-Period, Single-sequence, Drug-drug Interaction Study in Healthy Subjects to Assess the Effect of Cenicriviroc on the Pharmacokinetics (PK) of HMG-CoA Reductase Inhibitors [Rosuvastatin (ROS), Atorvastatin (ATO) and Simvastatin (SIM)], Caffeine and Digoxin

ELIGIBILITY:
Inclusion Criteria:

* Be informed of the nature of the study and have provided written informed voluntary consent.
* Have a BMI ≥ 18.0 and ≤ 35.0 kg/m2.
* Be in good general health with no clinically relevant abnormalities based on medical history, physical examination, clinical laboratory evaluations (clinical chemistry, hematology, urinalysis), and 12-lead ECG that, in the opinion of the Investigator, would affect subject safety.
* Be able to communicate effectively with the Investigator and other study center personnel and agree to comply with the study procedures and restrictions.

Exclusion Criteria:

* Any disease or condition that might affect drug absorption, metabolism, or excretion, or clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease, as determined by the Investigator and, if necessary, the Sponsor's Medical Monitor.
* History of stomach or intestinal surgery, except for fully healed appendectomy and/or cholecystectomy which will be allowed.
* Clinically significant illness or clinically significant surgery within 4 weeks before the administration of study medication.
* History of GERD, heartburn, or nausea more than once a month, or any similar symptoms requiring the regular use of antacids, or any use of H2 histamine blockers or proton-pump inhibitors over the past 3 months.
* History of achlorhydria, pernicious anemia, or peptic ulcers over the past 6 months.
* Known or suspected hypersensitivity or allergic reaction to any of the components of CVC, ROS, ATO, SIM, Digoxin or Caffeine tablets.
* History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin.
* If female, is pregnant or breast feeding, or has a positive pregnancy test result prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2016-02-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment of ROS, ATO and Digoxin alone and in the presence of CVC, as measured by maximum plasma concentration (Cmax) | Days 1 and 13
Pharmacokinetic Assessment of SIM alone and in the presence of CVC, as measured by maximum plasma concentration (Cmax) | Days 1 and 12
Pharmacokinetic Assessment of Caffeine alone and in the presence of CVC, as measured by maximum plasma concentration (Cmax) | Days 1 and 13
Pharmacokinetic Assessment of ROS, ATO and Digoxin alone and in the presence of CVC, as measured by minimum plasma concentration (Cmin) | Days 1 and 13
Pharmacokinetic Assessment of ROS, ATO and Digoxin alone and in the presence of CVC, as measured by area under the plasma concentration-time curve (AUC) | Days 1 and 13
Pharmacokinetic Assessment of SIM alone and in the presence of CVC, as measured by minimum plasma concentration (Cmin) | Days 1 and 12
Pharmacokinetic Assessment of SIM alone and in the presence of CVC, as measured by area under the plasma concentration-time curve (AUC) | Days 1 and 12
Pharmacokinetic Assessment of Caffeine alone and in the presence of CVC, as measured by minimum plasma concentration (Cmin) | Days 1 and 13
Pharmacokinetic Assessment of Caffeine alone and in the presence of CVC, as measured by area under the plasma concentration-time curve (AUC) | Days 1 and 13

SECONDARY OUTCOMES:
Evaluation of Adverse Events | 23 days
  Evaluate adverse events
Changes from Baseline in Clinical Laboratory Tests | Baseline and 23 days
  Evaluate changes from baseline in clinical laboratory tests including serum chemistry, and hematology
Changes from Baseline in 12-lead ECGs | Baseline and 23 days
  Evaluate changes from baseline in 12-lead ECGs
Changes from Baseline in Vital Signs | Baseline and 23 days
  Evaluate changes from baseline in vital signs, including blood pressure and pulse rate
Changes from Baseline in Physical Examinations | Baseline and 23 days
  Evaluate changes from baseline in physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Millie Gottwald, PharmD, Study Director — Tobira Therapeutics, Inc.
Locations (1):
- Miami, Florida, United States